CLINICAL TRIAL: NCT04221620
Title: Effectiveness of EEG Neurofeedback in Pediatric Occupational Therapy to Improve Executive Functioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northern Arizona University (Other)
Collaborators: Kidabilities Occupational Therapy Clinic (Unknown)
Responsible Party: Principal Investigator, Lauren Hall, Doctor of Occupational Therapy, Northern Arizona University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: northernAU
Record Dates: First submitted 2019-12-12; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Executive Functioning; Pediatric ALL
Keywords: EEG neurofeedback; occupational therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: One single group of 30 pediatric participants will undergo 20 sessions of traditional occupational therapy services while receiving EEG neurofeedback within each session. Standardized assessment will be administered at the beginning of the session and at the end of 20 sessions to compare differences between executive functioning skills.
Masking Description: Co-PI Catherine Young will be completing all evaluations and de-indentification of study participants. I (Lauren Hall) will be working with the de-identified data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EEG neurofeedback (Experimental): All participants will receive 20 sessions of traditional occupational therapy services while receiving EEG neurofeedback.
  Interventions: Device: Zengar Electroencephalogram (EEG) Neurofeedback device

INTERVENTIONS:
Device: Zengar Electroencephalogram (EEG) Neurofeedback device — Electroencephalogram (EEG) Neurofeedback is a noninvasive way to allow the central nervous system to self regulate and calm the brain enough to allow the frontal cortex to function in an ideal state, which is the part of the brain that controls important functions including behavior, problem solving, memory, language, emotions, and judgment. EEG Neurofeedback is performed via a musical medley that lasts for about 34 minutes, with baseline numbers taken at the beginning and after the music finishes. During this time, the participant will wear headphones, sensory clips on the ears (3 total), and two sensors on their head while receiving traditional occupational therapy services.

SUMMARY:
EEG Neurofeedback is a noninvasive way that allows the central nervous system to self regulate and the frontal cortex to be accessed through quieting of the limbic system at the subcortical level. Currently there is limited research in regards to the implications of EEG Neurofeedback, however, the investigators of this study have been using EEG Neurofeedback as a passive modality in the treatment of various pediatric clients with a variety of diagnoses and disorders. The purpose of this study is to determine whether or not EEG neurofeedback is effective in improving executive functioning skills in pediatric, school aged children as a modality in traditional occupational therapy services. The investigators hypothesize that EEG neurofeedback will assist with improved sensory gating abilities, therefore allowing for higher levels of cognition and awareness due to increased opportunities for the brain to regulate itself.

DETAILED DESCRIPTION:
Electroencephalogram (EEG) Neurofeedback is a noninvasive way to allow the central nervous system to self regulate and calm the brain enough to allow the frontal cortex to function in an ideal state, which is the part of the brain that controls important functions including behavior, problem solving, memory, language, emotions, and judgment. There is limited research in regards to the use of EEG Neurofeedback, however, occupational therapists Cat Young and Lauren Hall have been using EEG Neurofeedback alongside traditional therapy as 'background noise' with pediatric clients. These therapists have observed children experience steady increases in speech and language abilities, self-care tasks such as becoming potty trained, and better abilities to understand self-regulation of emotions with EEG Neurofeedback when used together with traditional occupational therapy services. EEG Neurofeedback is performed via a musical medley that lasts for about 34 minutes, with baseline numbers taken at the beginning and after the music finishes. During this time, the participant will wear headphones, sensory clips on the ears (3 total), and two sensors on their head.

The purpose of this study is to test the effectiveness of EEG Neurofeedback in improving executive functioning skills in pediatric school aged children. The investigators hypothesize is that the EEG Neurofeedback will allow the body to filter out unnecessary information and white noise to focus on the task at hand, and therefore access higher levels of cognition and awareness by helping the brain to regulate itself. This study does not require additional time outside of the therapy session. Some of these clients already received treatment in therapy. The purpose of this consent form is to use the data gained from the client's BRIEF-2 scores and therapy sessions to test effectiveness of this device.

Furthermore, the purpose of the study is to determine potential benefits of using EEG Neurofeedback alongside traditional occupational therapy in improving executive functioning skills in school aged children. Requirements include children who experience impairments based on scores of potentially clinically elevated or clinically elevated levels on the Behavior Rating Inventory of Executive Function 2, or the BRIEF-2. This assessment is considered the gold standard for testing executive functioning and has over 1000 peer reviewed articles. At time of evaluation, the parent(s) or legal caregiver(s) will be given one (1) BRIEF-2 parental rating scale, which will take an average of 10-15 minutes to complete. Each question will be answered via a three point scale for whether they see the specific behavior often, sometimes, or never. Potential benefits include improved ability to stay on task, organize and complete tasks. There is minimal risk associated with the use of EEG Neurofeedback. Children might experience discomfort with the sensors placed on their head and attached to their ears. Some children might initially feel uncomfortable with the experience of being a relaxed alert state if they are prone to being in heightened alert states.

ELIGIBILITY:
Inclusion Criteria:

* school aged children: ages 6 to 18 years old.
* score of 4 out of 9 on the BRIEF-2 assessment, indicating a potentially clinically elevated or clinically elevated need for therapeutic intervention

Exclusion Criteria:

* score of 3 or less of the 9 categories on the BRIEF
* ratings that are equal to or higher than 7 on the inconsistency scale (indicating parent/caregiver bias)
* age requirements not met

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Executive functioning improvements | minimum 20 weeks, up to 8 months
  Executive functioning improvements as indicated by improved scores on the Behavior Rating Inventory of Executive Functioning second edition, or BRIEF-2, at the end of 20 sessions when EEG neurofeedback was utilized. The BRIEF-2 is considered the gold standard for testing executive functioning and has over 1000 peer reviewed articles. It utilizes three different scoring sub-sections- typical, potentially clinically elevated. or clinically elevated. Participants in this study must score within the potentially clinically elevated or clinically elevated levels to qualify. Ideally, moving up one section to typical range or potentially elevated range would demonstrate positive study results.

CONTACTS AND LOCATIONS:
Locations (1):
- Kidabilities Occupational Therapy, Prescott, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Currently no plans to make individual participant data available. If plans change, all information will be de-identifiable and unable to be traced to specific participants.